CLINICAL TRIAL: NCT05080517
Title: What Are the Factors for Maintaining and Stopping of Accompanying Citizens? Do Personality Traits of Accompanying Citizens Appear to Influence These Factors?
Acronym: SPICES_MIX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0259 (SPICES_MIX)
Record Dates: First submitted 2021-09-30; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2017, cardiovascular diseases (CVDs) were the leading cause of death worldwide. Most cardiovascular diseases can be prevented by changing risk behaviors.

CVDs are distributed within a population along a socio-economic gradient. This is true within a country, but also between countries with different income levels. People living in a high-income country have better CVD health status than those living in a low-income country.

Several studies have shown that community-based primary prevention of cardiovascular disease can be effective. Other studies have shown that champions positively influence the implementation of health promotion strategies at the community level. These champions are people in the community who contribute to the implementation of new health programs by involving their local networks.

The SPICES project (Scaling-up Packages of Intervention for Cardiovascular disease prevention in selected sites in Europe and Sub-Saharan Africa) is an international study that aims to implement and evaluate a community-based cardiovascular disease prevention and control program. It involves 5 low, middle and high income countries, including populations in urban, semi-rural and rural areas. The study focused on four sets of interventions: health promotion, cardiovascular risk profiling, management and self-management and follow-up.

In France, the territory of Central West Brittany (CWB) was chosen to participate in the SPICES project because of the vulnerability of its population to cardiovascular disease.

It is in this context that a type 1 hybrid study is being set up in the CWB territory as part of the SPICES project.

For the quantitative part of the protocol (NCT03886064), a randomized controlled trial took place simultaneously to evaluate the effectiveness of a behavior change program led by community champions. Resident volunteers were selected based on their non-laboratory Interheart score. Those with a moderate risk were included in the trial. They were then distributed at random to an intervention group and a control group. The control group received minimal counseling. Those in the intervention group were brought together in support groups, with follow-up by champions.

In a type 1 hybrid trial, qualitative data on implementation are gathered.

This qualitative study will seek understand why participants in the SPICES project staying and/or stopping, from the point of view of champions A qualitative approach using semi-structured interviews and focus groups was used. The objective is to explore maintaining and/or stopping participants in the SPICES project, from the point of view of champions

ELIGIBILITY:
Inclusion Criteria :

* Patient over 18 years of age ;
* Have followed the training to the accompaniment proposed by the research team of SPICES ;
* Have signed the accompanying person's ethics charter co-created by the champions' research team.

Exclusion Criteria :

* Refusal of a champion to participate in the qualitative study ;
* Patients under judicial protection (guardianship, curatorship, ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The champions recruited in the SPICES study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Factors for maintaining or stopping | Day 1
  Evaluation of the factors or maintaining or stopping of accompanying citizens through semi-directed interviews. This is not a scale but an interview where feelings are evoked. No score.

SECONDARY OUTCOMES:
Perceived personality traits | Day 1
  Explore the correlations between the identified factors and the personality traits of the champions. The major personality traits of the accompanying citizens will be evaluated according to the Big Five Inventory 10 questionnaire (BFI-10). The BFI-10 is a 10-item scale measuring the Big Five personality traits Extraversion, Agreeableness, Conscientiousness, Emotional Stability, and Openness. The scale was developed based on the 44-item Big Five Inventory (BFI-44; John, Donahue, & Kentle, 1991; Rammstedt, 1997) and designed for contexts in which respondents' time is severely limited.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Jean-Yves Le Reste, Lanmeur, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion.